CLINICAL TRIAL: NCT05297994
Title: Trial of the Reactogenicity, Safety and Immunogenicity of the Flu-M Vaccine Manufactured by FSUE SPbSRIVS FMBA vs. the Vaxigrip® Inactivated Influenza Split Vaccine Manufactured by Sanofi Pasteur, France, in Volunteers Aged 18-60 Years
Brief Title: Trial of the Reactogenicity, Safety and Immunogenicity of the Flu-M Vaccine Manufactured by FSUE SPbSRIVS FMBA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Petersburg Research Institute of Vaccines and Sera (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FMV-VGIR-II-001/16
Record Dates: First submitted 2021-10-11; First posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2021-10

CONDITIONS: Influenza
Keywords: influenza; flu; vaccine; Flu-M
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flu-M (Experimental): 200 volunteers were vaccinated with the Flu-M inactivated split influenza vaccine with a preservative
  Interventions: Biological: Flu-M [Inactivated split influenza vaccine]
- Vaxigrip (Active Comparator): 200 volunteers were vaccinated with the Vaxigrip® inactivated split influenza vaccine
  Interventions: Biological: Inactivated influenza split vaccine

INTERVENTIONS:
Biological: Flu-M [Inactivated split influenza vaccine] — solution for intramuscular injection, 0.5 ml
  Arms: Flu-M
Biological: Inactivated influenza split vaccine — solution for intramuscular injection, 0.5 ml
  Arms: Vaxigrip

SUMMARY:
To trial the reactogenicity, safety and immunogenicity of the Flu-M inactivated split influenza vaccine in volunteers aged 18-60 years

DETAILED DESCRIPTION:
All subjects will be followed up for 21 days post-randomization. The subjects will further be assessed at 2 days, 7 days, 21 days following the booster vaccination. Blood samples will be collected for reactogenicity and safety and immunogenicity assessments before injection and 21 days after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent of the volunteers to participate in the clinical trial;
* Healthy volunteers (men and women) aged 18-60 years;
* Volunteers able to fulfill requirements of the protocol (fill out the patient's diary, come to follow-up visits);
* If the participant is female, she was required to have negative pregnancy test results and use contraceptives throughout the follow-up period (complete contraception of women of reproductive period)

Exclusion Criteria:

* Allergic reactions to chicken protein or any previous influenza vaccination;
* Leukemia, cancer or a positive reaction to human immunodeficiency virus infection, hepatitis B and C, syphilis in the past medical history;
* Volunteers who received immunoglobulin or blood products within the last 3 months before the trial;
* Guillain-Barré syndrome (acute polyneuropathy) in the medical history;
* Long-term use (more than 14 days) of immunosuppressants or other immunomodulatory drugs for 6 months prior to the trial.
* Any confirmed or suspected immunosuppressive or immunodeficiency condition;
* Respiratory, cardiovascular failure, impaired liver or kidney function found during a physical examination or laboratory tests during Visit 1;
* Severe birth defects or serious chronic diseases, including any clinically significant chronic diseases of lungs, kidneys, cardiovascular, nervous system, psychiatric diseases or metabolic disorders, confirmed by medical history or objective examination;
* Being (or having been) a patient of a tuberculosis dispensary and/or narcological dispensary and/or neuropsychiatric dispensary;
* acute infectious and/or non-infectious diseases at the time of inclusion in the trial;
* Exacerbation of chronic diseases;
* chronic alcohol abuse and/or use of drugs in the past history;
* Pregnancy and lactation;
* Participation in another clinical trial within the last 3 months;
* Immunization with influenza vaccines in the last 6 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2016-10-24 (Actual); Primary Completion 2016-12-12 (Actual); Study Completion 2017-03-09 (Actual)

PRIMARY OUTCOMES:
Severity of observed local reactions and their relationship with the vaccination | days 1-21 post-vaccination
  % of patients with:
  • Pain at the injection site at pressing Measurement tool: 4-point scale: 0 - none, 1 - mild, 2 - moderate, 3 - severe. Unit of measure: % of symptomatic patients at each severity
Severity of observed local reactions and their relationship with the vaccination | days 1-21 post-vaccination
  % of patients with:
  • Hyperemia; Measurement tool: 4-point scale: 0 - none, 1 - mild, 2 - moderate, 3 - severe. Unit of measure: % of symptomatic patients at each severity
Severity of observed local reactions and their relationship with the vaccination | days 1-21 post-vaccination
  % of patients with:
  • Infiltrate Measurement tool: 4-point scale: 0 - none, 1 - mild, 2 - moderate, 3 - severe. Unit of measure: % of symptomatic patients at each severity
Severity of observed local reactions and their relationship with the vaccination | days 1-21 post-vaccination
  % of patients with:
  • Swelling Measurement tool: 4-point scale: 0 - none, 1 - mild, 2 - moderate, 3 - severe. Unit of measure: % of symptomatic patients at each severity
Severity of observed system reactions and their relationship with the vaccination | days 1-21 post-vaccination
  % of patients with:
  • Fever Measurement tool: 4-point scale: 0 - none (≤ 37°С), 1 - mild (> 37°С - ≤ 37.5°С), 2 - moderate (> 37.6°С - ≤ 38.5°С), 3 - severe (> 38.6°С).
  Unit of measure: % of symptomatic patients at each severity
Severity of observed system reactions and their relationship with the vaccination | days 1-21 post-vaccination
  % of patients with:
  • Chills Measurement tool: 4-point scale: 0 - none, 1 - mild, 2 - moderate, 3 - severe. Unit of measure: % of symptomatic patients at each severity
Severity of observed system reactions and their relationship with the vaccination | days 1-21 post-vaccination
  % of patients with:
  • Increased sweating Measurement tool: 4-point scale: 0 - none, 1 - mild, 2 - moderate, 3 - severe. Unit of measure: % of symptomatic patients at each severity
Results of assessment of heart rate (HR) | days 1-21 post-vaccination
  The measurement of HR at each visit of the trial site by the volunteer
Results of assessment of systolic and diastolic blood pressure (BP) | days 1-21 post-vaccination
  The measurement of systolic and diastolic BP at each visit of the trial site by the volunteer
Results of biochemical blood tests | days 3, 7 and 21
  * ALT (U/L)
  * AST (U/L)
  * Alkaline phosphatase (U/L)
Results of biochemical blood tests | days 3, 7 and 21
  Bilirubin total (µmol/l)
Results of biochemical blood tests | days 3, 7 and 21
  Total protein (g/l)
Results of biochemical blood tests | days 3, 7 and 21
  C-reactive protein (mg/l)
Results of biochemical blood tests | days 3, 7 and 21
  * Urea (mmol/l)
  * Glucose (mmol/l)
  * Creatinine (mmol/l)
Results of complete blood counts | days 3, 7 and 21
  Erythrocytes (10^12/L)
Results of complete blood counts | days 3, 7 and 21
  Hemoglobin (g/L)
Results of complete blood counts | days 3, 7 and 21
  Erythrocyte sedimentation reaction (ESR) (mm/h)
Results of complete blood counts | days 3, 7 and 21
  Leukocytes, (х 10^9/L)
  Leukocytic formula:
  Stab neutrophils, % Segmented neutrophils (%) Eosinophils, (%) Basophils, (%) Lymphocytes, (%) Monocytes, (%)
Results of complete blood counts | days 3, 7 and 21
  Platelets, (х 10^9/L)
Incidence of AEs associated with the vaccination | days 1-21 post-vaccination
Incidence of SAEs associated with the vaccination | days 1-21 post-vaccination

CONTACTS AND LOCATIONS:
Locations (3):
- Russia (3):
  - Infection Center, Novosibirsk
  - Perm State Medical University named after Academician E. A. Wagner, Perm
  - Research Institute of Influenza, Saint Petersburg